CLINICAL TRIAL: NCT06803589
Title: Low-dose Growth Hormone for the Treatment of Gastroparesis
Brief Title: Growth Hormone for the Treatment of Gastroparesis
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Tisha N. Lunsford, GI and Hepatology Consultant, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24-003183
Record Dates: First submitted 2025-01-27; First posted 2025-01-31 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Gastroparesis
MeSH Terms: conditions — Gastroparesis | interventions — Growth Hormone; somapacitan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment Group (Experimental): Patients with Gastroparesis
  Interventions: Drug: Growth Hormone

INTERVENTIONS:
Drug: Growth Hormone — Subjects will receive growth hormone, Sogroya (Somapacitan-beco injections) via weekly injections for 12 weeks.
  For males, the fixed dose will be 0.2 mg/day, 1.5 mg per week
  For females, the fixed dose will be 0.3 mg/day, 2.1 mg per week
  Other Names: Sogroya (Somapacitan-beco injections)

SUMMARY:
The purpose of this study is to determine whether treatment with Growth Hormone results in symptomatic improvement in patients with gastroparesis.

ELIGIBILITY:
Inclusion Criteria:

* Symptoms > 6 months that have not responded satisfactorily to standard treatment.
* For gastroparesis: Gastroparesis Cardinal Symptom Index (GCSI) score of >21

Exclusion Criteria:

* Known history of GH deficiency, hypothalamic or pituitary disease
* Diabetes
* Prior use of GH therapy
* Age-adjusted low serum IGF1
* Women on oral estrogen therapy6
* Pregnancy or nursing
* History of malignant solid tumors
* Obesity (BMI > 30)History of coronary and thromboembolic diseases.
* History of sarcoidosis
* History of pituitary surgery
* History of thyroid nodules.
* Any other condition, which in the opinion of the investigator would impede compliance or hinder completion of the study.
* Failure to give informed consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-10-22 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Gastroparesis Cardinal Symptom Index (GCSI) | Baseline, 4 weeks, 8 weeks, 12 weeks, 14 weeks
  The Gastroparesis Cardinal Symptom Index (GCSI) is a questionnaire that assesses the severity of gastroparesis symptoms of: nausea, early satiety, postprandial fullness, and upper abdominal pain. Scores range from 0-none to 4-very severe.

SECONDARY OUTCOMES:
Complete Spontaneous Bowel Movements (CSBMs) | Baseline, 4 weeks, 8 weeks, 12 weeks, 14 weeks
  Number of bowel movements, without the aid of laxatives, after which the patient has the sensation of complete defecation.
Gastrointestinal Patient Reported Outcomes Measurement Information System (GI- PROMIS) | Baseline, 4 weeks, 8 weeks, 12 weeks, 14 weeks
  The Gastrointestinal Patient Reported Outcomes Measurement Information System (GI-PROMIS) scale assess 8 domains: gastroesophageal reflux, disrupted swallowing, diarrhea, bowel incontinence/soilage, nausea and vomiting, constipation, belly pain, and gas/bloat/flatulence. Scores are scaled so that an average healthy person would score 50 points. A higher score indicates worse gastrointestinal symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Tisha Lunsford, Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic, Phoenix, Arizona
  - Mayo Clinic in Arizona, Scottsdale, Arizona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials/cls-20574789